CLINICAL TRIAL: NCT00932841
Title: The Use of VSL#3 in Irritable Bowel Syndrome in Children
Acronym: VSL#3
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: PI has re-located. PI terminated FDA IND # and closed study.
Sponsor: Dayton Children's Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Sonia Michail, MD, Principal Investigator, Dayton Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 04-007; R21AT003400-01A2 (NIH)
Record Dates: First submitted 2009-07-02; First posted 2009-07-03 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- VSL#3 90 billion bacteria (Active Comparator)
  Interventions: Drug: VSL#3 90 billion bacteria
- VSL#3 900 billion bacteria (Active Comparator)
  Interventions: Drug: VSL#3 900 billion bacteria

INTERVENTIONS:
Other: Placebo — One packet PO daily x 8 weeks.
  Other Names: VSL#3
  Arms: Placebo
Drug: VSL#3 900 billion bacteria — One packet PO daily, x 8 weeks
  Other Names: VSL#3
  Arms: VSL#3 900 billion bacteria
Drug: VSL#3 90 billion bacteria — One packet PO daily, x 8 weeks.
  Other Names: VSL#3
  Arms: VSL#3 90 billion bacteria

SUMMARY:
The goal of this study is to determine whether the oral administration of the probiotic VSL#3 under randomized, placebo-controlled conditions will improve symptoms of irritable bowel syndrome in children, safely.

DETAILED DESCRIPTION:
Determine the safety and efficacy of different doses of VSL#3 in the treatment of children with irritable bowel syndrome: Children will be recruited from the pediatric gastroenterology clinic at The Children's Medical Center in Dayton, Ohio. Eighty four children will be enrolled in this controlled, double-blinded, randomized study. All children will have had a prior evaluation by a pediatric gastroenterologist who has diagnosed these patients with irritable bowel syndrome and excluded organic disease as a cause of the child's abdominal pain.

ELIGIBILITY:
Inclusion Criteria:

* All children should fulfill Rome ll criteria for IBS.
* Organic disease has been excluded.
* Age 13-18 years.
* Have active symptoms for at least 2 weeks prior to randomization. A minimum of 4.0 on the 7-point Likert scale for the two weeks prior to randomization on the GSRS-IBS composite pain score will be required.
* Diarrhea predominant IBS: Diarrhea is defined as increased stool frequency more than 3 times daily or change in form to loose or watery stools.

Exclusion Criteria:

* Children not fulfilling the inclusion criteria.
* Children receiving medication for the treatment of irritable bowel syndrome within 2 weeks of randomization.
* Children receiving antibiotic therapy or other probiotic agents within 4 weeks of randomization.
* Children receiving other medication known to cause abdominal pain.
* Children diagnosed with any of the following GI disorders: IBD (Crohn's disease or UC), Celiac disease, Gastroparesis, abdominal adhesions, Gastrointestinal perforation, Gastrointestinal obstruction and/or stricture, chronic or recurrent pancreatitis.
* Children who had undergone previous abdominal surgery (with the exception of uncomplicated appendectomy or cholecystectomy greater than or equal to 6 months prior to enrollment).
* Children with a history of any disease that may affect bowel motility such as diabetes mellitus, or poorly controlled hypo/hyperthyroidism.
* Children with immune deficiency, on immune-suppressants, or have active psychiatric, neurological, metabolic, renal, hepatic, infectious, hematological, cardiovascular or pulmonary disease.
* Children with a history of malignancy.
* Pregnancy.
* Children with history of allergy to maize or probiotics.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2008-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
The Gastrointestinal Symptom Rating Scale | 8 weeks

SECONDARY OUTCOMES:
Coddington life events questionnaire | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Michail, MD, Principal Investigator — Wright State University, Children's Medical Center of Dayton
Locations (1):
- Children's Medical Center of Dayton, Dayton, Ohio, United States

REFERENCES:
- [Background] APLEY J, NAISH N. Recurrent abdominal pains: a field survey of 1,000 school children. Arch Dis Child. 1958 Apr;33(168):165-70. doi: 10.1136/adc.33.168.165. No abstract available. PMID 13534750
- [Background] Everhart JE, Renault PF. Irritable bowel syndrome in office-based practice in the United States. Gastroenterology. 1991 Apr;100(4):998-1005. doi: 10.1016/0016-5085(91)90275-p. PMID 2001837
- [Background] Hamm LR, Sorrells SC, Harding JP, Northcutt AR, Heath AT, Kapke GF, Hunt CM, Mangel AW. Additional investigations fail to alter the diagnosis of irritable bowel syndrome in subjects fulfilling the Rome criteria. Am J Gastroenterol. 1999 May;94(5):1279-82. doi: 10.1111/j.1572-0241.1999.01077.x. PMID 10235207
- [Background] King TS, Elia M, Hunter JO. Abnormal colonic fermentation in irritable bowel syndrome. Lancet. 1998 Oct 10;352(9135):1187-9. doi: 10.1016/s0140-6736(98)02146-1. PMID 9777836
- [Background] Bengmark S. Ecological control of the gastrointestinal tract. The role of probiotic flora. Gut. 1998 Jan;42(1):2-7. doi: 10.1136/gut.42.1.2. No abstract available. PMID 9505873
- [Background] Nobaek S, Johansson ML, Molin G, Ahrne S, Jeppsson B. Alteration of intestinal microflora is associated with reduction in abdominal bloating and pain in patients with irritable bowel syndrome. Am J Gastroenterol. 2000 May;95(5):1231-8. doi: 10.1111/j.1572-0241.2000.02015.x. PMID 10811333
- [Background] Svedlund J, Sjodin I, Dotevall G. GSRS--a clinical rating scale for gastrointestinal symptoms in patients with irritable bowel syndrome and peptic ulcer disease. Dig Dis Sci. 1988 Feb;33(2):129-34. doi: 10.1007/BF01535722. PMID 3123181
- [Background] Balsari A, Ceccarelli A, Dubini F, Fesce E, Poli G. The fecal microbial population in the irritable bowel syndrome. Microbiologica. 1982 Jul;5(3):185-94. PMID 7121297